CLINICAL TRIAL: NCT05067153
Title: Thromboprophylaxis in Oesophageal Cancer Patients - A Randomized, Controlled Trial
Brief Title: Thromboprophylaxis in Oesophageal Cancer Patients
Acronym: TOP-RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-001335-24
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Esophageal Neoplasms; Thrombosis; Thromboembolism
Keywords: Esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Thrombosis; Thromboembolism | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial with one intervention group and one control group.
Masking Description: No masking due to ethical considerations. Primary outcome is biochemical.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group (n=50, anticipated) receives 30 days postoperative treatment with 5000 IE LMWH daily.
  Interventions: Drug: Fragmin 5000 UNT in 0.2 ML Prefilled Syringe
- Control (Active Comparator): Control group (n=50, anticipated) receives standard 10 days postoperative treatment with 5000 IE LMWH daily.
  Interventions: Drug: Fragmin 5000 UNT in 0.2 ML Prefilled Syringe

INTERVENTIONS:
Drug: Fragmin 5000 UNT in 0.2 ML Prefilled Syringe — 30 days postoperative prophylactic treatment.
  Other Names: Low Molecular Weight Heparin

SUMMARY:
The purpose of the study is to examine the efficacy and safety of prolonged thromboprophylactic treatment with Fragmin® in oesophageal cancer patients undergoing intended curative surgery.

DETAILED DESCRIPTION:
Hypotheses

1. The intervention group of oesophageal cancer patients, who receive prolonged thromboprophylaxis with Fragmin® has a lower VTE risk, expressed by a lower prothrombin fragment F1+2, 30 days after surgery than the control group, who receive Fragmin® for 10 days.
2. The intervention group does not demonstrate an increased bleeding tendency compared with the control group.

Primary endpoint The primary endpoint is the difference in prothrombin fragment F1+2 30 days after surgery between the intervention and the control group.

Secondary and safety endpoints The secondary endpoints are incidence of bleeding, VTE and mortality 30 days and one year after surgery.

Study design

The study is comprised of three specific objectives, presented in three work packages (WP):

* WP1: Randomization of 100 oesophageal cancer patients undergoing intended curative surgery to either a 10 or 30-day prophylactic LMWH-regime.
* WP2: Investigation of the coagulation in the WP1 population. The aim is to substantially improve understanding of the coagulation pathophysiology and the mechanisms behind the increased thromboembolic risk in oesophageal cancer patients.
* WP3: The lectin pathway complement proteins are suspected to play a role in the increased risk of thrombosis in cancer. We aim to examine this further by measuring complement protein levels in the WP1 population and investigate if there is a correlation between complement levels and changes in the coagulation.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer located in oesophagus and/or cardia.
2. Candidate for intended curative surgery.
3. Age > 18 years.

Exclusion Criteria:

1. Known inherited bleeding disorder.
2. Unable to provide informed consent.
3. Arterial or venous thromboembolic events within the last three months.
4. On-going anticoagulant treatment (Vitamin K antagonists or direct oral anticoagulants).
5. Pregnant or has given birth within the last three months.
6. Known allergy to the trial drug Dalteparin (Fragmin®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Prothrombin fragment F1+2 | 30 days after surgery.
  Difference in prothrombin fragment F1+2 between the intervention and the control group.

SECONDARY OUTCOMES:
Bleeding | 30 days after surgery.
  Incidence of bleeding
Venous thromboembolic events | 30 days and one year after surgery
  Incidence of venous thromboembolic events
Mortality | 30 days and one year after surgery
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Mette Hvas, MD, Principal Investigator — University of Aarhus
Locations (1):
- Thrombosis and Haemostasis Research Unit, Department for Clinical Biochemistry, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gyldenholm T, Madsen N, Katballe N, Kjaer DW, Christensen TD, Hvas AM. Patients Undergoing Oesophageal Cancer Surgery Do Not Have Impaired Haemostasis. Clin Appl Thromb Hemost. 2025 Jan-Dec;31:10760296251327587. doi: 10.1177/10760296251327587. Epub 2025 Mar 17. PMID 40095681
- [Derived] Gyldenholm T, Madsen N, Katballe N, Kjaer DW, Christensen TD, Hvas AM. Thromboprophylaxis in oesophageal cancer patients-a study protocol for a randomised, controlled trial (TOP-RCT). Trials. 2024 Sep 6;25(1):591. doi: 10.1186/s13063-024-08408-y. PMID 39242497